CLINICAL TRIAL: NCT04509778
Title: Develop a Psychosis Risk Calculator for Chinese Mental Health Servises
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, Associate Professor, Shanghai Mental Health Center
Other Study IDs: 16CR3016A
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Clinical High-risk
Keywords: calculator; conversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SHARP: ShangHai At Risk for Psychosis
  Interventions: Other: routine clinical treatment

INTERVENTIONS:
Other: routine clinical treatment — Participants will be informed that this is not a treatment study and it involves naturalistic follow-up without any extra intervention. They will otherwise follow the routine clinical treatment procedure.

SUMMARY:
This project will use the collected clinical and biological information of high-risk groups, use embedded computer chips, and use big data background analysis system to comprehensively evaluate the risk of high-risk groups, and build a mental illness risk estimator completely relying on the sample data of Chinese population and with independent intellectual property rights.

The calculator function and the risk calculation standard verified by the model can obtain the risk degree of each patient's progress to psychosis in the next two years. This calculator will play an important role in the prevention and treatment of psychosis.

DETAILED DESCRIPTION:
Severe mental disorders, mainly schizophrenia (SZ), affect 16 million Chinese population. At present, due to the lack of effective techniques and standards for early risk identification, the intervention opportunity for prevention and optimal efficacy is often missed.

In previous cohort studies , it has been found that this clinical high-risk(CHR) population can be effectively identified before its onset. Since 2011, the project team has been relying on the ShangHai At Risk for Psychosis Program, 300 CHRs were enrolled in the clinic through screening and diagnostic interview. The baseline clinical and event-related EEG indicators of this cohort were collected. The cohort was followed up for 2 years, with a follow-up completion rate of nearly 90%, it was found that the clinical outcome of high-risk groups was nearly one third, and the proportion of patients would be converted to schizophrenia within 2 years. This conversion rate is very consistent with the results of cohort studies of other large high-risk groups in the world. In view of this conversion ratio, many countries, such as the United States, have begun to use the baseline information to build prediction models, so as to form a psychiatric prediction tool.

After 5 years of accumulation, the project team has sufficient data to build a psychosis risk prediction model suitable for Chinese people, truly realize the goal of early diagnosis and treatment, and further support with the integration of key identification technologies and big data calculation.

ELIGIBILITY:
Inclusion Criteria:

* be aged 14 to 45-year-old;
* have had at least 6-years of primary education;
* be drug-naïve;
* be understanding the survey, be willing to enrol in the study and sign the informed consent;
* Through the Structured Interview for Prodromal Syndromes/Scale of Prodromal Symptoms (SIPS/SOPS), the participants should meet the Criteria of Prodromal Syndrome. Participants should fulfil at least one of the prodromal syndrome criteria: (1) brief intermittent psychotic syndrome, (2) attenuated positive symptom syndrome, or (3) genetic risk and deterioration syndrome.

Exclusion Criteria:

* Through the Mini-International Neuropsychiatric Interview (MINI), Axis I mental disorders such as schizophrenia, affective disorders, and anxiety spectrum disorders will be excluded;
* Acute or chronic renal failure; liver cirrhosis or active liver diseases;
* Abnormal laboratory tests results judged by the researchers to be clinically significant and considered to affect the efficacy of the test drugs or the safety of the subjects;
* Severe or unstable physical diseases, including: neurological disorders (delirium, dementia, stroke, epilepsy, migraine, etc.), congestive heart failure, angina pectoris, myocardial infarction, arrhythmia, hypertension (including untreated or uncontrolled hypertension), malignant tumours, immune compromise, and blood glucose above 12 mmol/L;
* Alcohol abuse within 30 days, or alcohol or drug dependence within 6 months before the trial;
* Pregnant or lactating women, or women in childbearing age who are positive in urine human chorionic gonadotropin test, or men and women who do not take effective contraceptive measures or plan for pregnancy within 3 months after the initiation of the trial;
* Stroke within the last month;
* Participating in any clinical trial within 30 days before the baseline;
* Other situations judged by the investigators not to be suitable for the clinical trial.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Help-seeking first-visit participants will be consecutively recruited from the Shanghai Psychotherapy and Psychological Counselling Centre at the Shanghai Mental Health Centre. They will be screened for eligibility by their clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Conversion to psychosis | 4 weeks
  It will be determined using the criteria for the Presence of Psychotic Symptoms from SIPS. Specifically, the conversion will be defined by the presence of level 6 positive symptoms (the rating "6" refers to severe and psychotic symptoms) identified as either dangerous, disorganised, or occurring at least one hour a day on average, over four days a week for at least 16 hours.
Poor function | 4 weeks
  It will be determined by GAF score. Specifically, poor function outcome is defined as the GAF score of less than 60 at the follow-up point.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code